CLINICAL TRIAL: NCT05271682
Title: A Phase I Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of the FHND6091 in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study Evaluating Safety, Tolerability and Clinical Activity of FHND6091 in Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Chia Tai Fenghai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LWY20071C
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1: 0.4 mg (Experimental): FHND6091, 0.4 mg, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091
- Part 1: 0.8 mg (Experimental): FHND6091, 0.8 mg, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091
- Part 1: 1.4 mg (Experimental): FHND6091, 1.4 mg, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091
- Part 1: 2.0 mg (Experimental): FHND6091, 2.0 mg, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091
- Part 1: 2.8 mg (Experimental): FHND6091, 2.8 mg, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091
- Part 1: 3.6 mg (Experimental): FHND6091, 3.6 mg, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091
- Part 2: lower dose expansion (Experimental): FHND6091, a lower dose, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091
- Part 2: MTD pr MTD-1 dose expansion (Experimental): FHND6091, MTD or MTD-1 dose, capsules, orally, once weekly on Days 1, 8, and 15 of a 28-day cycle in the dose escalation period
  Interventions: Drug: FHND6091

INTERVENTIONS:
Drug: FHND6091 — FHND6091 capsules

SUMMARY:
This is a phase I, first in human, single arm, open label study that will assess safety, tolerability and clinical activity of FHND6091 when taken orally on a weekly dosing schedule by patients with relapsed and refractory multiple myeloma (RRMM).The study will consist of two parts: dose escalation (Part 1) and dose expansion (Part 2).The dose escalation (Part 1) of the study will evaluate the safety and tolerability of FHND6091 using a dose escalation scheme to establish a maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D). And the dose expansion (Part B) of the study will further evaluate the safety, pharmacokinetics (PK)/ pharmacodynamics (PD), and efficacy of FHND6091 at two selected dose levels to characterize the safety, tolerability and efficacy of FHND6091.

A total of 40 evaluable participants will be enrolled in the study. The participants receiving treatment in part 1 and part 2 may continue combination treatment for a total of up to 12 cycles. After 12 cycles of therapy, the participants will continue treatment until the occurrence of PD, intolerable AEs, consent withdrawal, death or end of study based on the judgement of investigator's assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent.
* Male or female patients 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
* Life expectancy of at least 12 weeks.
* Patients with multiple myeloma who have relapsed or refractory, intolerance or refuse treatment following at least 3 regimens or lines of therapy that must include an IMID (lenalidomide or thalidomide), a proteasome inhibitor (bortezomib) , a CD38-targeted mAbs and corticosteroids. Patients must have received transplant therapy or are not suitable for transplant.
* For Patients With Relapsed Refractory Multiple Myeloma must have measurable disease defined by at least 1 of the following 2 measurements: Serum M-protein ≥ 5 g/L, or Urine M-protein ≥ 200 mg/24 hours. For patients with serum free light chain as measurable disease: Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa to lambda free light chain ratio.
* Clinical laboratory values as specified below within 14 days before the first dose of study drug:

  1. Hemoglobin ≥ 75 g/L, Absolute neutrophil count ≥ 1.0 x 10E9/L and Platelet count ≥ 75 x 10E9/L without blood transfusion, EPO or G-CSF and other medical support for at least 14 days prior to receiving screening.
  2. Total bilirubin levels ≤ 2 x ULN, AST (SGOT) and ALT (SGPT) ≤ 2 x ULN.
  3. Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/minute as calculated by Cockcroft-Gault method.
  4. Corrected Serum Calcium ≤ ULN.
* For man and women of childbearing potential: agreement to remain abstinent or use contraception, during the treatment period (including treatment interruptions) and for at least 180 days after the last dose of FHND6091 was administered. Women of childbearing potential should be negative by serum pregnancy test within 7 days prior dosing.

Exclusion Criteria:

* Documented allergy to proteasome inhibitor or ；
* Patients with peripheral neuropathy ≥ Grade 2 or Grade 1 peripheral neuropathy with pain.
* Patients with diarrhea > Grade 1 (Increase of <4 stools per day over baseline; mild increase in ostomy output compared to baseline).
* Patients received chemotherapy, radiation therapy, targeted therapy, immunotherapy or other systemic anticancer therapy within 14 days prior FHND6091 treatment.
* Patients received ixazomib treatment within 5 elimination half-life prior first dose of FHND6091 treatment.
* Patients received allogeneic stem cell transplantation or autologous stem cell transplant with 12 weeks before screening.
* Patients with symptomatic brain metastases, leptomeningeal metastases or, spinal cord compression or central nervous system (CNS) injuries/abnormalities based on investigator judgement.
* Evidence of severe or uncontrolled systemic diseases (eg, unstable or uncompensated respiratory, hepatic or renal disease), or receive major surgery.
* Patients with unstable hypertension after drug treatment (SBP ≥140 mmHg, DBP ≥90 mmHg ) or heart failure, myocardial ischemia or myocardial infarction, unstable angina, arrhythmia (The corrected QT interval (Fridericia formula) interval (QTcF) > 470 msec for females and > 450 msec for men in electrocardiogram (ECG)).
* Patients with active, or a history of immunodeficiency, including HIV positive or other acquired and congenital immunodeficiency diseases, or a history of solid organ transplant.
* Patients with a history of other serious underlying diseases, such as: a, history of a clear neurological or psychiatric disorder, including epilepsy or dementia. b, HBV surface antigen positivity (subjects with documented laboratory evidence of HBV clearance may be enrolled) or positive HCV antibody. c, presence of infection requiring systemic treatment.
* Systemic treatment with strong inhibitors of of CYP3A4 or strong CYP3A4 inducers within 5 elimination half-life prior first dose of FHND6091 treatment.
* Patients have not recovered (ie, ≤ Grade 1 toxicity by CTCAE 5.0) from the reversible effects of prior antineoplastic therapy (except for alopecia )
* Patients with other malignancy；
* Treatment with any investigational products within 28 days before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Treatment-Emergent Adverse Events and Serious Adverse Events | Baseline to 28 days after first dose of FHND6091 administration
  An Adverse Event is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
  A Serious Adverse Event (SAE) was any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.

SECONDARY OUTCOMES:
Complete Response/Stringent Complete Response (CR/sCR) Rate | Baseline to 12 months after first dose of FHND6091 administration
  CR/sCR to FHND6091, according to international myeloma working group (IMWG) criteria
Rate of Very Good Partial Response (VGPR) or Better | Baseline to 12 months after first dose of FHND6091 administration
  VGPR to FHND6091, according to international myeloma working group (IMWG) criteria
Partial Response (PR) | Baseline to 12 months after first dose of FHND6091 administration
  PR to FHND6091, according to international myeloma working group (IMWG) criteria
Cmax: Maximum Observed Plasma Concentration for FHND6091 | Days 1 and 15 of Cycle 1 (each cycle is 28 days)
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve for FHND6091
Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for FHND6091 | Days 1 and 15 of Cycle 1 (each cycle is 28 days)
  Time to reach the maximum observed plasma concentration (Cmax), equal to time to Cmax
AUC(0-168): Area Under the Plasma Concentration-Time Curve From Time 0 to 168 Hours Postdose for FHND6091 | Days 1 and 15 of Cycle 1 (each cycle is 28 days)
  AUC(0-168) is a measure of the area under the plasma concentration-time curve over the dosing interval (tau) (AUC[0-tau]), where tau is the length of the dosing interval - 168 hours in this study)

CONTACTS AND LOCATIONS:
Overall Officials: Jianqin Mi, M.D., Principal Investigator — Ruijin Hospital
Locations (6):
- China (6):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Third Hosptial of Changsha, Changsha, Hunan
  - The Affilitated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Ruijin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No